CLINICAL TRIAL: NCT04175262
Title: Clinical Effectiveness of Second-Line Sunitinib Following Immune-oncologic (IO) Therapy in Patients With Metastatic Renal Cell Carcinoma in the International Metastatic Renal Cell Carcinoma Database (IMDC)
Brief Title: Clinical Outcomes For Patients With Metastatic Renal Cell Carcinoma (mRCC) Who Received Sunitinib After 1st Line Immune-oncology (IO) Treatments
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) (Other); Analysis Group, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181233
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Results first posted 2021-04-02 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Renal Cell Carcinoma (mRCC)
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with mRCC: Patients diagnosed with metastatic RCC receiving first line (1L) combination of IOs therapies followed by Sunitinib as a second line (2L) treatment
  Interventions: Drug: sunitinib

INTERVENTIONS:
Drug: sunitinib — Patients to receive sunitinib as second line therapy for mRCC

SUMMARY:
The study aims to assess clinical outcomes in mRCC patients treated with sunitinib in second-line following IO therapy in real world clinical practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

  * Diagnosed with mRCC
  * Received IO therapy as 1L therapy
  * Received sunitinib as 2L therapy
  * Age 18 years or over at the time of mRCC diagnosis
  * Actively treated at an IMDC clinical center (to avoid incomplete data)

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with diagnosis of mRCC who initiated sunitinib as 2nd line treatment
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6181233

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants included in this study, were diagnosed with metastatic renal cell carcinoma (mRCC), who were treated with sunitinib from 2014 to 2019, after first-line immune-oncologic therapy.
Pre-assignment Details: In this study, data for participants was collected retrospectively through the international mRCC database consortium (IMDC) database. Data was collected and analyzed during study duration of approximately 4 months.
Groups:
- Sunitinib Following Immune-oncologic Therapy: Participants with mRCC who received sunitinib as second line therapy from 2014 to 2019 after first line immune-oncologic therapy in real world clinical practices were included in this study.
Period: Overall Study
Arm/Group | Sunitinib Following Immune-oncologic Therapy
Started | 102
Completed | 102
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data was collected and analyzed in this study.
Arm/Group | Sunitinib Following Immune-oncologic Therapy
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 78
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 54
  Race: Non-White | 48
Prior Nephrectomy Status [Count of Participants; unit: Participants] — Here, number of participants with their previous nephrectomy status as "Yes" or "No" are reported.
  Participants
    Yes | 78
    No | 24
Histology Type [Count of Participants; unit: Participants] — Here, number of participants with histology type as "Clear cell" or "Non-clear cell" are reported. Population: Here 'number analyzed" signifies participants evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 88
    Clear cell | 81
    Non-clear cell | 7
Metastatic Sites [Count of Participants; unit: Participants] — Here, number of participants are classified according to number of metastatic sites. Population: Here 'number analyzed" signifies participants evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 83
    Greater than (>) 1 | 77
    1 | 6
Site of Metastases [Count of Participants; unit: Participants] — Here, number of participants are classified according to type of metastatic sites. Population: Here 'Number analyzed" signifies participants evaluable for this baseline measure.
  Participants
    Lung: number analyzed (Participants) | 83
    Lung | 36
    Lymph nodes: number analyzed (Participants) | 83
    Lymph nodes | 26
    Bone: number analyzed (Participants) | 83
    Bone | 22
    Liver: number analyzed (Participants) | 83
    Liver | 12
    Brain: number analyzed (Participants) | 83
    Brain | 8
    Adrenal gland: number analyzed (Participants) | 83
    Adrenal gland | 7
    Pancreas: number analyzed (Participants) | 83
    Pancreas | 5
    Other (Soft tissues, kidney, pleura, pelvis, spleen, peritoneum, and perineal fat): number analyzed (Participants) | 83
    Other (Soft tissues, kidney, pleura, pelvis, spleen, peritoneum, and perineal fat) | 21
Participants According to Time From RCC Diagnosis to First Line Therapy [Count of Participants; unit: Participants] — Here, number of participants are classified according to duration of RCC diagnosis to first line therapy.
  Participants
    Less than (<) 1 year | 67
    Greater than or equal to (>= 1) year | 35
Karnofsky Performance Status (KPS) [Count of Participants; unit: Participants] — KPS is a standard way of measuring the ability of participants with cancer to perform ordinary tasks. KPS scores range from 0 percent (%) (dead) to 100% (normal, no complaints). A higher score means the participant is better able to carry out daily activities. Here, number of participants are classified with KPS score of <80% and >=80%. Population: Here 'number analyzed" signifies participants evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 91
    < 80% | 23
    >= 80% | 68
Hemoglobin Level [Count of Participants; unit: Participants] — Here, number of participants are classified with hemoglobin level < lower limit normal (LLN) and >= LLN. Population: Here 'number analyzed" signifies participants evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 91
    < LLN | 57
    >=LLN | 34
Serum Corrected Calcium Level [Count of Participants; unit: Participants] — Here, number of participants are classified with serum corrected calcium level > upper limit normal (ULN) and <= ULN. Population: Here 'number analyzed" signifies participants evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 83
    > ULN | 5
    Less than or equal to (<=) ULN | 78
Neutrophil Count [Count of Participants; unit: Participants] — Here, number of participants are classified with neutrophil count > ULN and <= ULN. Population: Here 'number analyzed" signifies participants evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 90
    > ULN | 22
    <= ULN | 68
Platelets Count [Count of Participants; unit: Participants] — Here, number of participants are classified with platelets count > ULN and <= ULN. Population: Here 'number analyzed" signifies participants evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 91
    > ULN | 17
    <= ULN | 74

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) After Initiation of Second Line Sunitinib Therapy
Description: Overall survival was defined as the time (in months) from second line sunitinib initiation to death. Participants were censored at their date of last follow-up. Kaplan-Meier method was used for analysis.
Time Frame: From the date of initiation of second line sunitinib to the date of death or censored date, up to a maximum of approximately 5.5 years (from the data collected and observed retrospectively for approximately 4 months)
Population: Analysis population included all eligible participants whose data was collected and analyzed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib Following Immune-oncologic Therapy
Number analyzed (Participants) | 102
Months | 15.6 [9.8 to 21.7]

2. Primary Outcome: Time to Treatment Discontinuation (TTD) of Second Line Sunitinib Therapy
Description: TTD was defined as the time (in months) between initiation of second line sunitinib therapy and discontinuation of therapy for any reason including progression, death, and toxicity. Participants were censored at their date of last follow-up. As per response evaluation criteria in solid tumors (RECIST) 1.1 criteria: disease progression was at least a 20% increase in sum of diameters of target lesions, taking as a reference smallest sum on treatment, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm), or the appearance of at least 1 new lesion. Unequivocal progression of existing non-target lesions. Kaplan-Meier method was used for analysis.
Time Frame: From the date of initiation of second line sunitinib to discontinuation or censored date, up to a maximum of approximately 5.5 years (from the data collected and observed retrospectively for approximately 4 months)
Population: Analysis population included all eligible participants whose data was collected and analyzed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib Following Immune-oncologic Therapy
Number analyzed (Participants) | 102
Months | 5.4 [4.2 to 7.2]

3. Primary Outcome: Time to Treatment Discontinuation (TTD) of First Line Immune-Oncologic Therapy
Description: TTD was defined as the time (in months) between initiation of first line Immune-Oncologic therapy and discontinuation of therapy for any reason including progression, death, and toxicity. Participants were censored at their date of last follow-up. As per RECIST 1.1 criteria: disease progression was at least a 20% increase in sum of diameters of target lesions, taking as a reference smallest sum on treatment, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of at least 1 new lesion. Unequivocal progression of existing non-target lesions. Kaplan-Meier method was used for analysis.
Time Frame: From the initiation of immune-oncologic therapy to discontinuation of immune-oncologic therapy (approximately up to 2 years)
Population: Analysis population included all eligible participants whose data was collected and analyzed in this study.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Sunitinib Following Immune-oncologic Therapy
Number analyzed (Participants) | 102
Months | 7.4 (8.8)

4. Primary Outcome: Number of Participants Classified According to Reasons for Second-Line Sunitinib Treatment Discontinuation
Description: Reasons for treatment discontinuation included disease progression, death, toxicity and other reasons including urosepsis, nausea, vomiting, diarrhea, comorbidity, and other unspecified. As per RECIST v1.1. criteria, disease progression was at least a 20% increase in sum of diameters of target lesions, taking as a reference smallest sum on treatment, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of at least 1 new lesion. Unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 2
Population: Analysis population included all eligible participants whose data was collected and analyzed in this study. Here, "Overall Number of Participants Analyzed" signifies participants who discontinued second line sunitinib treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib Following Immune-oncologic Therapy
Number analyzed (Participants) | 58
Participants
  Disease progression | 28
  Toxicity | 17
  Death | 3
  Disease progression and Toxicity | 1
  Disease progression and Death | 1
  Other (urosepsis, nausea, vomiting, diarrhea, comorbidity, and other unspecified) | 8

5. Primary Outcome: Objective Response Rate (ORR) After Initiation of Second Line Sunitinib Therapy
Description: The objective response rate was defined as the percentage of participants with partial response (PR) and complete response (CR). As per RECIST 1.1 criteria: CR = disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalisation of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis); PR = at least 30% decrease in sum of diameters of target lesions taking as reference baseline sum diameters.
Time Frame: From the date of initiation of second line sunitinib to the date of PR and CR or censored date, up to a maximum of approximately 5.5 years (from the data collected and observed retrospectively for approximately 4 months)
Population: Analysis population included all eligible participants whose data was collected and analyzed in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sunitinib Following Immune-oncologic Therapy
Number analyzed (Participants) | 102
Percentage of participants | 22.5 [12.6 to 32.5]

6. Primary Outcome: Percentage of Participants With Progressive Disease (PD) After Initiation of Second Line Sunitinib Therapy
Description: Progressive disease (PD) was defined as an increase in visible disease. According to RECIST 1.1; PD = at least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on the study. This includes the baseline sum if that is the smallest on study. In addition to the relative increase of 20%, the sum also demonstrated an absolute increase of at least 5 mm or the appearance of at least 1 new lesion. Unequivocal progression of existing non-target lesions.
Time Frame: From the date of initiation of second line sunitinib to occurrence of disease progression, up to a maximum of approximately 5.5 years (from the data collected and observed retrospectively for approximately 4 months)
Population: Analysis population included all eligible participants whose data was collected and analyzed in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sunitinib Following Immune-oncologic Therapy
Number analyzed (Participants) | 102
Percentage of participants | 43.7 [31.8 to 55.5]

7. Primary Outcome: Percentage of Participants With Stable Disease (SD) After Initiation of Second Line Sunitinib Therapy
Description: Stable disease was defined as no change in size of visible disease. According to RECIST 1.1, stable disease: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease , taking as reference the smallest sum diameters while on study; PD = at least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on the study. This includes the baseline sum if that is the smallest on study. In addition to the relative increase of 20%, the sum also demonstrated an absolute increase of at least 5 mm or the appearance of at least 1 new lesion. Unequivocal progression of existing non-target lesions. PR = at least 30% decrease in sum of diameters of target lesions taking as reference baseline sum diameters.
Time Frame: From the date of initiation of second line sunitinib to the date stable disease or censored date, up to a maximum of approximately 5.5 years (from the data collected and observed retrospectively for approximately 4 months)
Population: Analysis population included all eligible participants whose data was collected and analyzed in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sunitinib Following Immune-oncologic Therapy
Number analyzed (Participants) | 102
Percentage of participants | 33.8 [22.5 to 45.1]

8. Primary Outcome: Time From First Line Immune-Oncologic Therapy Discontinuation to Initiation of Second Line Sunitinib Therapy
Time Frame: From the discontinuation of immune-oncologic therapy to the initiation of sunitinib therapy (approximately up to 2 years)
Population: Analysis population included all eligible participants whose data was collected and analyzed in this study.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Sunitinib Following Immune-oncologic Therapy
Number analyzed (Participants) | 102
Months | 3.1 (6.2)

9. Primary Outcome: Number of Participants Classified According to Reasons for First-Line Immune-Oncologic Treatment Discontinuation
Description: Reasons for treatment discontinuation included disease progression, toxicity and other reasons including itchiness, mouth dryness, comorbidity, and other unspecified. As per RECIST 1.1 criteria: disease progression was at least a 20% increase in sum of diameters of target lesions, taking as a reference smallest sum on treatment, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of at least 1 new lesion. Unequivocal progression of existing non-target lesions.
Time Frame: From the date of initiation of first line Immune-Oncologic to discontinuation or follow-up (approximately up to 2 years)
Population: Analysis population included all eligible participants whose data was collected and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib Following Immune-oncologic Therapy
Number analyzed (Participants) | 102
Participants
  Disease progression | 53
  Toxicity | 23
  Disease progression and Toxicity | 1
  Other (itchiness, mouth dryness, comorbidity, and other unspecified) | 25

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events not collected during the study
Description: Due to the nature of claims database from which data were queried, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) would not meet, hence safety data was not planned to be collected and reported.
Arm/Group | Sunitinib Following Immune-oncologic Therapy
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT04175262/Prot_SAP_000.pdf